CLINICAL TRIAL: NCT06694051
Title: Application of Phototherapeutic Keratectomy Mode to Mark the Axis of Astigmatism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2024055
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ptk-group (Experimental)
  Interventions: Procedure: marking
- limbus-group (No Intervention)

INTERVENTIONS:
Procedure: marking — axis marking
  Arms: ptk-group

SUMMARY:
Corneal refractive surgery is an effective way to correct refractive error. Modern corneal refractive surgery for the correction of myopia or hyperopia can achieve or close to the expected goal, but to eliminate astigmatism is always one of the major problems of corneal refractive surgery. The key point in the correction of astigmatism is that as a vector parameter, astigmatism has both magnitude and direction. The angle error may be caused by the rotation of the patient's head position and the involuntary rotation of eyes. Phototherapeutic keratectomy can precisely cut the corneal tissue, and is often used in clinic to remove corneal scars or repair corneal surface morphology. In this study, the excimer laser therapeutic keratectomy mode was used to achieve accurate marking of the axis of astigmatism by setting the treatment laser parameters. With the help of the static cyclotorsion of the eye, the precise treatment of astigmatism could realize.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old

Exclusion Criteria:

* ocular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
refraction | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China